CLINICAL TRIAL: NCT01243580
Title: An Open-Label Study to Evaluate Pharmacokinetic Profile of Agile TCDS AG200-15 and to Compare Exposure to Ethinyl Estradiol to Oral Contraceptive (Orthocyclen®) in Healthy Female Volunteers
Brief Title: AG200-15 Transdermal Contraceptive Delivery System (TCDS) of Levonorgestrel and Ethinyl Estradiol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agile Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ATI-CL14
Record Dates: First submitted 2010-11-16; First posted 2010-11-18 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Healthy
Keywords: PK and safety; Pharmacokinetic profile (PK) and safety
MeSH Terms: interventions — Moxifloxacin; Contraceptives, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ortho-Cyclen® (Active Comparator): Ortho-Cyclen® is a comparator drug intervention
  Interventions: Drug: Ortho-Cyclen
- AG200-15 (Experimental): AG200-15 is an investigational transdermal contraceptive delivery system that is a drug intervention
  Interventions: Drug: AG200-15

INTERVENTIONS:
Drug: Ortho-Cyclen — Ortho-Cyclen is an oral contraceptive containing 35 µg of EE and 250 µg of norgestimate (NGM) in a 21 - 7 day regimen.
  Other Names: oral contraceptive
  Arms: Ortho-Cyclen®
Drug: AG200-15 — AG200-15 is a transdermal contraceptive delivery system delivering 100 - 120 mcg of LNG and 25 - 30 mcg EE
  Other Names: transdermal contraception
  Arms: AG200-15

SUMMARY:
Pharmacokinetics and safety of AG200-15 over two consecutive cycles of therapy will be evaluated.

DETAILED DESCRIPTION:
This is an open-label study comprised of two parts. Part I is a single-arm, run-in cycle with AG200-15 administered to all subjects as a 21-7 day regimen (three consecutive weeks of patch wear followed by a patch-free week).

Part II employs crossover design with subjects randomly assigned to one of the two treatment sequences. Each sequence will include AG200-15 and oral contraceptive (Ortho-Cyclen®) as described below: Sequence 1: AG200-15 (Period 1) followed by oral contraceptive, Ortho-Cyclen® (Period 2); Sequence 2: Oral contraceptive, Ortho-Cyclen® (Period 1) followed by AG200-15 (Period 2) Both AG200-15 and Ortho-Cyclen® will be administered as 21-7 day regimen (three consecutive weeks of drug-taking followed by a drug-free week). Duration of each treatment Period is 28 days (one cycle of therapy).

ELIGIBILITY:
Inclusion Criteria:

* Healthy women, ages 18-45
* Body mass index (BMI) ≥18 and ≤32, and weight ≥ 110 lbs.
* Willing to use a non-hormonal method of contraception if at risk of pregnancy, OR have already undergone previous bilateral tubal ligation or hysterectomy
* Willing to refrain from use of alcohol and grapefruit juice from 48 hours prior until completion of each treatment period

Exclusion Criteria:

* Known or suspected pregnancy;
* Lactating women
* Significant skin reaction to transdermal preparations or sensitivity to surgical / medical tape
* Any disease that may worsen under hormonal treatment (cardiovascular, liver, metabolic)
* Use of other contraceptive methods than study medication
* Smokers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Garner, MD, MPH, Study Director — Agile Therapeutics
Locations (1):
- Miami, Florida, United States

REFERENCES:
- [Derived] Archer DF, Stanczyk FZ, Rubin A, Foegh M. Ethinyl estradiol and levonorgestrel pharmacokinetics with a low-dose transdermal contraceptive delivery system, AG200-15: a randomized controlled trial. Contraception. 2012 Jun;85(6):595-601. doi: 10.1016/j.contraception.2011.10.006. Epub 2011 Nov 30. PMID 22133660

RESULTS

PARTICIPANT FLOW:
Groups:
- AG200-15/Ortho-Cyclen®: AG200-15 transdermal contraceptive delivery system, delivering 25-30 mcg ethinyl estradiol/ 100-120 mcg levonorgestrel per day, was applied weekly for 3 consecutive weeks and was removed on the 4th week for a patch free week. This regimen occurred for Cycles 1 and 2. For cycle 3, Ortho-Cyclen® containing 250 mcg norgestimate and 35 mcg ethinyl estradiol was taken daily for 21 days followed by a drug free interval of 7 days.
- Ortho-Cyclen®/AG200-15: AG200-15 transdermal contraceptive delivery system, delivering 25-30 mcg ethinyl estradiol and 100-120 mcg levonorgestrel per day, was applied for 3 consecutive weeks and removed on the 4th week for a patch free week. This regimen occurred for Cycle 1 and Cycle 3. Ortho-Cyclen®, containing 250 mcg norgestimate and 35 mcg ethinyl estradiol, was taken daily for 21 days followed by a drug free interval of 7 days for Cycle 2.
Period: Overall Study
Arm/Group | AG200-15/Ortho-Cyclen® | Ortho-Cyclen®/AG200-15
Started | 18 | 18
Completed | 18 | 16
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- AG200-15/Ortho-Cyclen®: Subject applied AG200-15 in cycle 1. Subjects applied AG200-15 (Cycle 2) followed by oral contraceptive, Ortho-Cyclen® (Cycle 3)
- Ortho-Cyclen® /AG200-15: Subject applied AG200-15 in cycle 1. Subjects received Ortho-Cyclen® (Cycle 2) followed by AG200-15 (Cycle 3).
- Total: Total of all reporting groups
Arm/Group | AG200-15/Ortho-Cyclen® | Ortho-Cyclen® /AG200-15 | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (5.85) | 36.2 (7.66) | 37 (6.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Comparative Evaluation of Ethinyl Estradiol (EE) Cmax Between AG200-15 and Ortho-Cyclen® in Week 1
Description: Comparative evaluation of ethinyl estradiol (EE) Cmax between AG200-15 and Ortho-Cyclen® in week 1 for cycle 2 and 3.
Time Frame: 3 months
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- AG200-15: AG200-15 is an investigational transdermal contraceptive delivery system that is a drug intervention
  AG200-15: AG200-15 is a transdermal contraceptive delivery system delivering 100 - 120 mcg of levonorgestrel (LNG) and 25 - 30 mcg EE
Arm/Group | Ortho-Cyclen® | AG200-15
Number analyzed (Participants) | 29 | 33
pg/ml | 135 (50.7) | 45.5 (24.0)
Statistical Analysis 1: Comparison: Ortho-Cyclen® vs AG200-15; Test type: Equivalence — Comparing Ortho-Cyclen to Ag200-15; p < 0.0001, ANOVA

2. Primary Outcome: Comparative Evaluation of EE Cmax Between AG200-15 and Ortho-Cyclen® in Week 3
Description: Comparative evaluation of EE Cmax between AG200-15 and Ortho-Cyclen® in week 3 for cycles 2 and 3.
Time Frame: 3 months
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Ortho-Cyclen® | AG200-15
Number analyzed (Participants) | 32 | 32
pg/ml | 131 (45.4) | 51.3 (17.3)
Statistical Analysis 1: Comparison: Ortho-Cyclen® vs AG200-15; Test type: Equivalence — Comparison of AG200-15 and Ortho-Cyclen; p < 0.0001, ANOVA

3. Primary Outcome: Comparative Evaluation of EE AUC(0-168hrs Post-first Dose) Between AG200-15 and Ortho-Cyclen® in Week 1
Description: Comparative evaluation of EE AUC (0-168hrs post-first dose) between AG200-15 and Ortho-Cyclen® in week 1 for cycles 2 and 3.
Time Frame: 3 months
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: ng.h/ml
Arm/Group | Ortho-Cyclen® | AG200-15
Number analyzed (Participants) | 29 | 32
ng.h/ml | 7.28 (2.66) | 5.06 (2.26)
Statistical Analysis 1: Comparison: Ortho-Cyclen® vs AG200-15; Test type: Equivalence — Comparison of AG200-15 and Ortho-Cyclen; p = 0.0001, ANOVA

4. Primary Outcome: Comparative Evaluation of EE AUC (0-168hrs Post-first Dose) Between AG200-15 and Ortho-Cyclen® in Week 3
Description: Comparative evaluation of EE AUC (0-168hrs post-first dose) between AG200-15 and Ortho-Cyclen® in week 3 for cycles 2 and 3.
Time Frame: 3 months
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: ng.h/ml
Arm/Group | Ortho-Cyclen® | AG200-15
Number analyzed (Participants) | 32 | 32
ng.h/ml | 6.97 (2.25) | 6.26 (2.46)
Statistical Analysis 1: Comparison: Ortho-Cyclen® vs AG200-15; Test type: Equivalence — Comparison of Ortho-Cylen and AG200-15; p = 0.0532, ANOVA

5. Primary Outcome: Comparative Evaluation of EE Css (1) Between AG200-15 and Ortho-Cyclen® in Week 1
Description: Comparative evaluation of EE Css (1) between AG200-15 and Ortho-Cyclen® in week 1 for cycles 2 and 3. For Ortho-Cyclen steady-state concentration calculated as average concentration at steady-state from the 24-hour trapezoidal AUC (AUC0-24h/24). For AG200-15 the average concentration within the 48-168 h time-interval was measured.
Time Frame: 3 months
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Ortho-Cyclen® | AG200-15
Number analyzed (Participants) | 32 | 32
pg/ml | 43.3 (15.8) | 31.4 (15.1)
Statistical Analysis 1: Comparison: Ortho-Cyclen® vs AG200-15; Test type: Equivalence — Comparison of Ortho-Cyclen and AG200-15; p = 0.0009, ANOVA

6. Primary Outcome: Comparative Evaluation of EE Css (1) Between AG200-15 and Ortho-Cyclen® in Week 3
Description: Comparative evaluation of EE Css (1) between AG200-15 and Ortho-Cyclen® in week 3 for cycles 2 and 3. For Ortho-Cyclen steady-state concentration calculated as average concentration at steady-state from the 24-hour trapezoidal AUC (AUC0-24h/24). For AG200-15 the average concentration within the 48-168 h time-interval was measured.
Time Frame: 3 months
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Ortho-Cyclen® | AG200-15
Number analyzed (Participants) | 32 | 32
pg/ml | 41.5 (13.4) | 35.7 (14.5)
Statistical Analysis 1: Comparison: Ortho-Cyclen® vs AG200-15; Test type: Equivalence — Comparison of Ortho-Cyclen and AG200-15; p = 0.0167, ANOVA

7. Primary Outcome: Comparative Evaluation of EE Css (2) Between AG200-15 and Ortho-Cyclen® in Week 1
Description: Comparative evaluation of EE Css (2) between AG200-15 and Ortho-Cyclen® in week 1 for cycles 2 and 3. For Ortho-Cyclen steady-state concentration calculated as average concentration at steady-state from the 24-hour trapezoidal AUC (AUC0-24h/24). For Ag200-15, the average concentration at steady-state calculated from trapezoidal AUC within the 48-168h time interval (AUC/time interval).
Time Frame: 3 months
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Ortho-Cyclen® | AG200-15
Number analyzed (Participants) | 32 | 32
pg/ml | 43.3 (15.8) | 32.0 (16.2)
Statistical Analysis 1: Comparison: Ortho-Cyclen® vs AG200-15; Test type: Equivalence — Comparison of Ortho-Cyclen and AG200-15; p = 0.0007, ANOVA

8. Primary Outcome: Comparative Evaluation of EE Css (2) Between AG200-15 and Ortho-Cyclen® in Week 3
Description: Comparative evaluation of EE Css (2) between AG200-15 and Ortho-Cyclen® in week 3 for cycles 2 and 3. For Ortho-Cyclen steady-state concentration calculated as average concentration at steady-state from the 24-hour trapezoidal AUC (AUC0-24h/24). For Ag200-15, the average concentration at steady-state calculated from trapezoidal AUC within the 48-168h time interval (AUC/time interval).
Time Frame: 3 months
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Ortho-Cyclen® | AG200-15
Number analyzed (Participants) | 32 | 32
pg/ml | 41.5 (13.4) | 35.7 (15.4)
Statistical Analysis 1: Comparison: Ortho-Cyclen® vs AG200-15; Test type: Equivalence — Comparison of Ortho-Cyclen and AG200-15; p = 0.0175, ANOVA

9. Primary Outcome: Comparative Evaluation of EE Css (3) Between AG200-15 and Ortho-Cyclen® in Week 1
Description: Comparative evaluation of EE Css (3) between AG200-15 and Ortho-Cyclen® in week 1 for cycles 2 and 3. For Ortho-Cyclen steady-state concentration calculated as average concentration at steady-state from the 24-hour trapezoidal AUC (AUC0-24h/24). For AG200-15, the average concentration at steady-state calculated from trapezoidal AUC within the 0-168h time interval (AUC/time interval).
Time Frame: 3 months
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Ortho-Cyclen® | AG200-15
Number analyzed (Participants) | 32 | 32
pg/ml | 43.3 (15.8) | 30.1 (13.4)
Statistical Analysis 1: Comparison: Ortho-Cyclen® vs AG200-15; Test type: Equivalence — Comparison of Ortho-Cyclen and AG200-15; p = 0.0001, ANOVA

10. Primary Outcome: Comparative Evaluation of EE Css (3) Between AG200-15 and Ortho-Cyclen® in Week 3
Description: Comparative evaluation of EE Css (3) between AG200-15 and Ortho-Cyclen® in week 3 for cycles 2 and 3. For Ortho-Cyclen steady-state concentration calculated as average concentration at steady-state from the 24-hour trapezoidal AUC (AUC0-24h/24). For AG200-15, the average concentration at steady-state calculated from trapezoidal AUC within the 0-168h time interval (AUC/time interval).
Time Frame: 3 months
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Ortho-Cyclen® | AG200-15
Number analyzed (Participants) | 32 | 32
pg/ml | 41.5 (13.4) | 37.3 (14.7)
Statistical Analysis 1: Comparison: Ortho-Cyclen® vs AG200-15; Test type: Equivalence — Comparison of Ortho-Cyclen and AG200-15; p = 0.0532, ANOVA

11. Primary Outcome: Evaluation of LNG Cmax Between AG200-15 in Week 1 and 3
Description: Evaluation of LNG Cmax Between AG200-15 in Week 1 and 3 for cycles 2 and 3.
Time Frame: 3 months
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | AG200-15
Number analyzed (Participants) | 33
pg/ml
  Week 1 | 1370 (908)
  Week 3 | 2400 (1140)

12. Primary Outcome: Evaluation of LNG AUC (0-168hrs Post-first Dose) Between AG200-15 in Week 1 and 3
Description: Evaluation of LNG AUC (0-168hrs post-first dose) Between AG200-15 in Week 1 and 3 for cycles 2 and 3.
Time Frame: 3 months
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: ng.h/ml
Arm/Group | AG200-15
Number analyzed (Participants) | 33
ng.h/ml
  Week 1 | 160 (88.9)
  Week 3 | 317 (159)

13. Primary Outcome: Evaluation of LNG Css (1) Between AG200-15 in Week 1 and 3
Description: Comparative evaluation of EE Css (1) between AG200-15 and Ortho-Cyclen® in week 1 for cycles 2 and 3. For Ortho-Cyclen, steady-state concentration calculated as average concentration at steady-state from the 24-hour trapezoidal AUC (AUC0-24h/24). For Ag200-15, the average concentration at steady-state calculated from trapezoidal AUC within the 48-168h time interval (AUC/time interval).
Time Frame: 3 months
Population: Primary PK population
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | AG200-15
Number analyzed (Participants) | 33
pg/ml
  Week 1 | 1060 (631)
  Week 3 | 1847 (930)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events were analyzed based on Organ System class.
Arm/Group | Ortho-Cyclen® | AG200-15
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/36
Other Adverse Events (participants affected / at risk) | 3/34 | 23/36
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ortho-Cyclen® (N=34) | AG200-15 (N=36)
Gastointestinal disorders (Gastrointestinal disorders) | 2 (2) | 6 (6)
General disorders and application site conditions (General disorders) | 1 (1) | 8 (8)
Infections and infestations (Infections and infestations) | 1 (1) | 3 (3)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscoloskeletal and conncetive tissue disoders (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nervous system disoders (Nervous system disorders) | 0 (0) | 17 (17)
Reproductive system and breast disoders (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Approval by Agile Therapeutics, Inc. of any publication, including oral presentations and abstracts, utilizing data or any information from the ATI-CL14 study is required prior to publication submission.